CLINICAL TRIAL: NCT00687154
Title: An Observational Study of the Development of Diabetic Macular Edema Following Scatter Laser Photocoagulation
Brief Title: Observational Study of DME Following Scatter Laser Photocoagulation
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Director, Jaeb Center for Health Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NEI-127; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Laser; macular edema; retinopathy; scatter photocoagulation
MeSH Terms: conditions — Macular Edema; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Sitting (Active Comparator): Subjects with (1) OCT central subfield thickness ≤ 299 microns and (2) early proliferative or severe nonproliferative diabetic retinopathy for which investigator intends to perform full scatter photocoagulation in 1 sitting
  Interventions: Procedure: Scatter Laser Photocoagulation in 1 Sitting
- 4 Sittings (Active Comparator): Subjects with (1) OCT central subfield thickness ≤ 299 microns and (2) early proliferative or severe nonproliferative diabetic retinopathy for which investigator intends to perform full scatter photocoagulation in 4 sittings.
  Interventions: Procedure: Scatter Laser Photocoagulation in 4 Sittings

INTERVENTIONS:
Procedure: Scatter Laser Photocoagulation in 1 Sitting — 1 sitting with a minimum of 1200 to a maximum of 1600 burns, with one burn width separation of burns and scatter extending from the peripheral arcades to beyond the equator.
  Other Names: PRP
  Arms: 1 Sitting
Procedure: Scatter Laser Photocoagulation in 4 Sittings — 4 sittings, each separated by four weeks (+4 days), with approximately 300 burns in each of the first two sittings and investigator judgment for number of burns for the third and fourth sittings as long as the total for the four sittings is between 1200 and 1600 burns.
  Other Names: PRP
  Arms: 4 Sittings

SUMMARY:
The development or worsening of macular edema following full scatter photocoagulation is a well recognized occurrence. However, there is limited literature in this regard.

The purpose of this study is to determine the incidence and extent of macular edema following scatter laser photocoagulation surgery using optical coherence tomography (OCT) in eyes without macular edema prior to scatter laser photocoagulation and to explore whether the incidence and extent of macular edema varies according to the number of sittings included in the treatment regimen.

Study eyes will receive one of two types of scatter photocoagulation with results compared through use of OCT and photography images, as well as visual acuity testing.

DETAILED DESCRIPTION:
Study eyes will receive scatter photocoagulation given by one of the following two regimens. To reduce selection bias, investigators will be required, prior to study initiation, to indicate which treatment (1 PRP sitting or 4 PRP sittings) they will administer. Only the selected treatment will be performed by a given investigator on study eyes.

* 1 sitting with a minimum of 1200 to a maximum of 1600 burns, with one burn width separation of burns and scatter extending from the peripheral arcades to beyond the equator.
* 4 sittings, each separated by four weeks (+4 days), with approximately 300 burns in each of the first two sittings and investigator judgment for number of burns for the third and fourth sittings as long as the total for the four sittings is between 1200 and 1600 burns.

Both of these regimens conform with usual clinical practice.

The study aims to enroll 150 eyes. At least 40 eyes will be enrolled with prior focal laser photocoagulation and at least 40 eyes without prior focal laser treatment. After enrollment of 80 eyes (40 with prior treatment and 40 without prior treatment), an interim analysis will be conducted so that focused enrollment strategies can be implemented if the analysis suggests that more subjects in a subgroup should be entered. Approximately half of the eyes will receive each scatter treatment regimen.

The following procedures will be done on the study eye at baseline and at each scheduled visit (except 8 and 12 weeks at which exam data are not collected) unless otherwise specified:

* OCT
* E-ETDRS visual acuity in both eyes (refraction in the study eye at baseline, 17 weeks, and 34 weeks)
* Fundus photographs (7-fields at baseline and 3-fields at 34 weeks only)
* Photographs to document the scatter photocoagulation (day of the first PRP sitting only)

ELIGIBILITY:
Inclusion Criteria: To be eligible, the following inclusion (1-4) and exclusion criteria (5-8) must be met:

1. Age >= 18 years

   • Patients <18 years old are not being included because there would be an insufficient number of patients <18 years old who would meet eligibility criteria for the study in order to be able to generalize the results to patients <18 years old or to provide informative data as to the effects of treatment in this age group.
2. Diagnosis of diabetes mellitus (type 1 or type 2)

   • Any one of the following will be considered to be sufficient evidence that diabetes is present:
   1. Current regular use of insulin for the treatment of diabetes
   2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   3. Documented diabetes by ADA and/or WHO criteria
3. At least one eye meets the study eye criteria listed in section 2.2.2.
4. Able and willing to provide informed consent.

   Exclusion Criteria: A patient is not eligible if any of the following exclusion criteria (5-8) are present:
5. History of chronic renal failure requiring dialysis or kidney transplant.
6. History of pancreatic transplant.
7. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

   • Patients in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
8. Patient is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 8 months.

The patient must have at least one eye meeting all of the inclusion criteria (a-d) and none of the exclusion criteria (e-k) listed below.

A patient can have only one study eye. If both eyes are eligible, the investigator at his/her discretion will select one to be the study eye.

The eligibility criteria for a study eye are as follows:

Inclusion

1. Presence of early proliferative or severe nonproliferative diabetic retinopathy for which investigator intends to perform full scatter photocoagulation in either one sitting or four sittings.
2. Central subfield thickness on OCT ≤ 299 microns. Note: Clinically significant macular edema is not an exclusion provided the central subfield is ≤299 microns.
3. Visual acuity 73 letters or greater (20/32 or better).
4. Media clarity, pupillary dilation, and patient cooperation sufficient to administer full scatter photocoagulation and obtain adequate fundus photographs and OCT.

   Exclusion
5. Prior scatter photocoagulation.
6. High risk (severe proliferative) retinopathy.
7. Presence of an ocular condition (other than diabetes) that, in the opinion of the investigator, might produce macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, significant vitreomacular interface disease, etc.).
8. Treatment for diabetic macular edema is planned.
9. History of any treatment for DME within prior 6 months, including focal/grid macular photocoagulation and corticosteroids by any route.
10. History of major ocular surgery (including cataract extraction, vitrectomy, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 8 months following enrollment.
11. History of YAG capsulotomy performed within 2 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Retinal thickening (measured with OCT) | 34 weeks

SECONDARY OUTCOMES:
Visual Acuity (measured with E-ETDRS) | 2 days, 4 weeks, 17, and 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J. Brucker, M.D., Study Chair — Scheie Eye Institute

REFERENCES:
- [Result] Diabetic Retinopathy Clinical Research Network; Brucker AJ, Qin H, Antoszyk AN, Beck RW, Bressler NM, Browning DJ, Elman MJ, Glassman AR, Gross JG, Kollman C, Wells JA 3rd. Observational study of the development of diabetic macular edema following panretinal (scatter) photocoagulation given in 1 or 4 sittings. Arch Ophthalmol. 2009 Feb;127(2):132-40. doi: 10.1001/archophthalmol.2008.565. PMID 19204228